CLINICAL TRIAL: NCT01832181
Title: Metformin in Women With Type 2 Diabetes in Pregnancy Kids Trial (MiTy Kids)
Brief Title: MiTy Kids (Metformin in Women With Type 2 Diabetes in Pregnancy Kids Trial)
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Research Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 10-0129-A
Record Dates: First submitted 2013-04-08; First posted 2013-04-15 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; MiTy; Metformin in Women; Type 2 Diabetes Pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Metformin
- Control

SUMMARY:
The prevalence of diabetes in pregnancy is rising in all maternal age groups. There is increasing evidence that in-utero exposure to maternal diabetes is associated with an increased risk of obesity and type 2 diabetes in children and adults. There is an urgent need to reduce these increasing rates of obesity and diabetes in subsequent generations.

The MiTy Trial (Metformin in Women with Type 2 Diabetes in Pregnancy Trial) is a CIHR-funded multi-centre, randomized controlled trial of women with type 2 diabetes in pregnancy (sample size n=500). The MiTy Trial is looking to determine the effect of the addition of metformin to a standard regimen of insulin in women with diabetes, on perinatal morbidity and mortality.

The MiTy Kids Trial is a follow-up to the MiTy Trial which will determine whether treatment with metformin during pregnancy in women with type 2 diabetes will lead to a reduction in adiposity and improvement in insulin resistance in the offspring of women with diabetes at 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Offspring of women with type 2 diabetes who participated (or are participating) in the MiTy trial.

Exclusion Criteria:

* Offspring with major congenital anomalies.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Offspring of women with type 2 diabetes who participated in the MiTy trial during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2013-04; Primary Completion 2021-04 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Adiposity in the offspring | 24 months
  Anthropometric measures: BMI and sum of skinfolds (triceps, subscapular, suprailiac and biceps).

SECONDARY OUTCOMES:
Sum of skinfolds in the offspring | 6, 12 and 24 months
  Triceps, subscapular, suprailiac and biceps.
Central to peripheral adiposity in the offspring | 6, 12 and 24 months
  Suprailiac to triceps skinfold ratio.
Weight gain, BMI and weight-for-length percentile change over time in critical early periods and overall in the offspring. | 3, 6, 12, 18 and 24 months
  Weight and length.
Overweight and obesity in the offspring | 3, 6, 12, 18 and 24 months
  BMI >85th percentile (overweight) and BMI >97th percentile (obesity) for age and gender from World Health Organization (WHO) growth charts.
Insulin resistance in the offspring | 24 months
  Fasting insulin, fasting insulin-to-glucose ratio, and the Homeostasis Model of Assessment - Insulin Resistance (HOMA-IR).
adipocytokine profile in the offspring | 24 months
  Adiponectin and leptin.

CONTACTS AND LOCATIONS:
Overall Officials: Denice Feig, MD, Principal Investigator — Mount Sinai Hospital, Toronto, Ontario, Canada
Locations (1):
- Dr. Denice Feig, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Feig DS, Sanchez JJ, Murphy KE, Asztalos E, Zinman B, Simmons D, Haqq AM, Fantus IG, Lipscombe L, Armson A, Barrett J, Donovan L, Karanicolas P, Tobin S, Mangoff K, Klein G, Jiang Y, Tomlinson G, Hamilton J; MiTy Kids Collaborative Group. Outcomes in children of women with type 2 diabetes exposed to metformin versus placebo during pregnancy (MiTy Kids): a 24-month follow-up of the MiTy randomised controlled trial. Lancet Diabetes Endocrinol. 2023 Mar;11(3):191-202. doi: 10.1016/S2213-8587(23)00004-9. Epub 2023 Feb 3. PMID 36746160